CLINICAL TRIAL: NCT04242316
Title: Effects of Mirror Therapy and Bilateral Arm Training on Hemiparetic Upper Extremity in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20121012008
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stroke; Hemiplegia
Keywords: Stroke; Mirror therapy; Bilateral arm training; Upper limb function
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Experimental): Patients performed customized bimanual upper limb exercises with a mirror. They can observe the mirror visual feedback of their non-paretic hand during the movements.
  Interventions: Behavioral: Mirror Therapy
- Bilateral arm training (Active Comparator): Patients performed customized bimanual upper limb exercises without a mirror.
  Interventions: Behavioral: Bilateral arm training

INTERVENTIONS:
Behavioral: Mirror Therapy — Patients performed customized bimanual upper limb exercises with graded level of difficulty based on the patient's individual levels of upper limb functioning according to the 7 levels of the FTHUE and each level consisted of 5 standardized table-top tasks. The patients practiced the movements with the unaffected hand (including the shoulder, elbow, wrist, and hand). While watching the reflection of the unaffected hand in the mirror, the patient was then asked to moving the affected hand at the same time to synchronize the movement with the reflection of the unaffected hand. If the patient was unable to move the hand, a therapist would passively assist the movement of the affected hand so as to synchronize it with the reflection of the unaffected hand.
  Arms: Mirror Therapy
Behavioral: Bilateral arm training — Patients performed customized bimanual upper limb exercises with graded level of difficulty based on the patient's individual levels of upper limb functioning according to the 7 levels of the FTHUE and each level consisted of 5 standardized table-top tasks, but without a mirror. The patients can take a direct view of their paretic hand.
  Arms: Bilateral arm training

SUMMARY:
The aim of this study included (1) to compare the effectiveness of mirror therapy (MT) and bimanual arm training (BAT) in improving motor and functional performance of hemiplegic upper extremity for adults with chronic stroke; (2) to examine whether recruitment of the mirror neurons, as reflected in mu rhythm suppression, mediates recognition of the mirror illusion in pre/post MT, as compared to BAT without a mirror in clients with chronic stroke, as compared to healthy participants.

DETAILED DESCRIPTION:
Mirror Therapy (MT) appeared to have beneficial effects on the recovery of distal function of the hemiplegic hand in the evidence recently, however, it is not known whether the incongruent visual feedback induced by mirror in bilateral arm training (BAT) is beneficial to the motor performance of upper extremity than without the mirror in patients with chronic stroke. This study aimed to compare the effectiveness of MT and bimanual arm training (BAT) in improving motor and functional performance of hemiplegic upper extremity for adults with chronic stroke. Participants with chronic stroke were recruited by convenience sampling from a convalescent hospital and self-help groups in the community in Hong Kong. Participants were randomly assigned to the MT group or BAT group and participated in a 6-week upper limb training programme which consisted of two 45-minute training sessions per week. Both kinds of training were equivalent to each other except that there was a mirror used in the MT group. Main outcome measures were upper extremity motor and functional tests, and grip strength. Participants were evaluated at baseline, post-treatment and 3-month follow-up. EEG was assessed before and after the training in a group of stroke patients and healthy controls, in order to evaluate the recruitment of the mirror neurons, as reflected in mu rhythm suppression.

ELIGIBILITY:
Inclusion Criteria:

1. neurological condition with unilateral hemiparesis;
2. a Functional Test of Hemiplegic Upper Extremity (FTHUE) score between levels 2 to 6;
3. chronic stroke with onset of neurological condition more than 6 months previously;
4. ability to understand and follow simple verbal instructions;
5. ability to participate in a therapy session lasting at least 30 minutes;
6. community ambulant with or without aids.

Exclusion Criteria:

Individuals with severe neglect and severe spasticity (Modified Ashworth Scale >3) would be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment (FMA) | Baseline
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Fugl-Meyer assessment (FMA) | After 6-week
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Fugl-Meyer assessment (FMA) | 3-month after the completion of training
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Action Research Arm Test (ARAT) | After 6-week
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Action Research Arm Test (ARAT) | 3-month after the completion of training
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Wolf Motor Function Test (WMFT) | Baseline
  WMFT assesses the functional limitation of upper limb after a neurological condition. This test evaluates both strength (2 items) and function-based task performance (15 items).
Wolf Motor Function Test (WMFT) | After 6-week
  WMFT assesses the functional limitation of upper limb after a neurological condition. This test evaluates both strength (2 items) and function-based task performance (15 items).
Wolf Motor Function Test (WMFT) | 3-month after the completion of training
  WMFT assesses the functional limitation of upper limb after a neurological condition. This test evaluates both strength (2 items) and function-based task performance (15 items).

OTHER OUTCOMES:
Mu rhythm suppression generated in the sensorimotor cortex | Baseline
  Electroencephalographical assessment for cortical activation induced by mirror visual feedback.
Mu rhythm suppression generated in the sensorimotor cortex | 6-week
  Electroencephalographical assessment for cortical activation induced by mirror visual feedback.

IPD SHARING:
Plan to Share IPD: No